CLINICAL TRIAL: NCT03858049
Title: Comparison of Crinone ® Versus Combination Medication for Luteal Phase Support on the Ongoing Pregnancy Rate of Frozen-thawed Cycle in Chinese Population a Randomized, Interventional, Open-label, Phase IV, Single Center, Pilot Study (ACCESS)
Brief Title: Efficacy and Safety of Crinone Versus Combination Medication (ACCESS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trend in LPS treatment tends to increase the dosage of progesterone in FET-HRT, this study was designed 5 years ago.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200113_0005
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Infertility
Keywords: Frozen-thawed embryo transfer; Infertility; Crinone; Duphaston; Chinese population
MeSH Terms: conditions — Infertility | interventions — Crinone; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crinone (Experimental): Participants received Crinone 8% (90 milligrams [mg] an intravaginal progesterone gel contained in a single use, one piece applicator) once daily in morning from the day of endometrial transformation (Day -5) until ongoing pregnancy was confirmed up to Day 63.
  Interventions: Drug: Crinone
- Crinone plus Duphaston (Experimental): Participants received Crinone 8% (90 mg an intravaginal progesterone gel contained in a single use, one piece applicator) once daily in morning followed by 10 mg of Duphaston tablet orally twice a day from the day of endometrial transformation (Day -5) until ongoing pregnancy was confirmed up to Day 63.
  Interventions: Drug: Crinone; Drug: Duphaston

INTERVENTIONS:
Drug: Crinone — Participants received Crinone 8% (90 milligrams [mg] an intravaginal progesterone gel contained in a single use, one piece applicator) once daily in morning from the day of endometrial transformation (Day -5) until ongoing pregnancy was confirmed up to Day 63.
Drug: Duphaston — Participants received 10 mg of Duphaston tablet orally twice a day from the day of endometrial transformation (Day -5) until ongoign pregnancy was confirmed up to Day 63.
  Arms: Crinone plus Duphaston

SUMMARY:
The study to compare to the efficacy and safety of Crinone versus combination medication in infertile women receive frozen-thawed embryo transfer (FET) in artificial cycles (AC).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

* Participants who will receive artificial frozen-thawed embryo transfer (FET) cycle study interventions
* Participants who have no more than two Day 5 embryos are planned to be transferred (follow the clinical practice of the study site)
* Participants have received estradiol valerate for no more than 20 days
* Participants have a transitional-endometrium of greater than or equal to 8 millimeter
* Participants have normal uterine cavity
* Participants can give signed informed consent
* Participants are willing to follow the study protocol and able to complete the study

Exclusion Criteria:

* Participants are willing to follow the study protocol and able to complete the study
* Participants with greater than or equal to three previously failed cycles of ET
* Participants with diseases that cannot tolerate pregnancy
* Hydrosalpinx
* Severe endometriosis (Endometriosis American Society for Reproductive Medicine (ASRM) criteria from 1996)
* Known hypersensitivity to progesterone, the excipients of Crinone and Duphaston Vaginal bleeding of unknown origin
* History of recurrent miscarriages
* Vaginitis
* Thromboembolic diseases (thrombophlebitis, thromboembolic disorder, or cerebral apoplexy) or participants with a history of these conditions
* Known or suspected progestogen-dependent neoplasm
* Participation in another clinical trial within the past 30 days
* Contraindications of both Crinone and Duphaston

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200113_0005
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Crinone® Plus Duphaston: Participants received Crinone 8% (90 mg an intravaginal progesterone gel contained in a single use, one piece applicator) once daily in morning followed by 10 mg of Duphaston tablet orally twice a day from the day of endometrial transformation (Day -5) until ongoing pregnancy was confirmed up to Day 63.
Period: Overall Study
Arm/Group | Crinone | Crinone® Plus Duphaston
Started | 86 | 86
Completed | 69 | 76
Not Completed | 17 | 10
Not completed — Adverse Event | 16 | 9
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population included all participants who received at least one dose of randomized study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crinone | Crinone® Plus Duphaston | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.84 (2.918) | 30.74 (3.163) | 30.79 (3.034)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 86 | 86 | 172
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy Rate
Description: Ongoing pregnancy was assessed by the presence of viable intra uterine fetus detected by ultrasound examination in 10-12 weeks of pregnancy (8 to 10 weeks after embryo transfer). Ongoing pregnancy rate is defined as the number of participants with ongoing pregnancy divided by the number of participants with embryo transfer (ET) multiplied by 100.
Time Frame: 8 to 10 weeks after embryo transfer
Population: ITT Population included all participants who received at least one dose of randomized study intervention. Here, "Number of participants analyzed" signified those participants who had embryo transferred.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 85 | 86
Percentage of participants | 18.8 [11.2 to 28.8] | 29.1 [19.8 to 39.9]

2. Secondary Outcome: Beta Human Chorionic Gonadotrophin (Beta-hCG) Positive Rate
Description: Beta-hCG positive rate defined as number of participants with positive beta-hCG divided by the number of participants with embryo transfer (ET) multiplied by 100.
Time Frame: 2 weeks after embryo transfer
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 85 | 86
Percentage of participants | 37.6 [27.4 to 48.8] | 43.0 [32.4 to 54.2]

3. Secondary Outcome: Implantation Rate
Description: Implantation rate was measured as the number of gestational sacs observed divided by the number of embryos transferred (ET) multiplied by 100.
Time Frame: 4-6 weeks after embryo transfer
Population: ITT Population included all participants who received at least one dose of randomized study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of gestational sacs per ET
Units Other Than Participants: embroys transferred
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 86 | 86
Number analyzed (embroys transferred) | 86 | 86
percentage of gestational sacs per ET | 20.9 [12.9 to 31.0] | 33.7 [23.9 to 44.7]

4. Secondary Outcome: Clinical Pregnancy Rate
Description: Clinical Pregnancy was defined as the pregnancy diagnosed by ultrasound of one or more gestational sacs or definitive clinical signs of pregnancy. Clinical pregnancy rate was measured as the number of participants with clinical pregnancy divided by number of participants with embryo transfer (ET) multiplied by 100.
Time Frame: 4-6 weeks after embryo transfer
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 85 | 86
Percentage of participants | 21.2 [13.1 to 31.4] | 33.7 [23.9 to 44.7]

5. Secondary Outcome: Early Abortion Rate
Description: Early abortion defined as the spontaneous loss of an intra-uterine pregnancy prior to 12 completed weeks of gestational age. Early abortion rate defined as the number of participants with early abortion divided by number of participants with clinical pregnancy multiplied by 100.
Time Frame: Time from embryo transfer to 12 weeks of pregnancy
Population: ITT Population included all participants who received at least one dose of randomized study intervention. Here, "Number of participants analyzed" signified those participants with clinical pregnancy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 18 | 29
Percentage of participants | 11.1 [1.4 to 34.7] | 13.8 [3.9 to 31.7]

6. Secondary Outcome: Luteal Phase Bleeding Rate
Description: Luteal Phase Bleeding defined as the onset of any bleeding after embryo transfer and prior to the pregnancy test. Luteal phase bleeding rate defined as the number of participants with Luteal phase bleeding divided by number of participants with embryo transfer (ET) multiplied by 100.
Time Frame: 2, 5 and 9 weeks after embryo transfer
Population: Safety analysis set included all participants who have received at least one dose of study intervention. Here, "Number of participants analyzed" signified those participants who had embryo transferred.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 85 | 86
Percentage of participants | 1.2 [0.0 to 6.4] | 3.5 [0.7 to 9.9]

7. Secondary Outcome: Vaginal Bleeding Rate
Description: Vaginal bleeding is defined as any bleeding recorded after a pregnancy test via serum Beta-Human Chorionic Gonadotrophin. Vaginal bleeding rate defined as the number of participants with vaginal bleeding divided by number of participants with embryo transfer (ET) multiplied by 100.
Time Frame: 5 and 9 weeks after embryo transfer
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Crinone | Crinone® Plus Duphaston
Number analyzed (Participants) | 85 | 86
Percentage of participants | 7.1 [2.6 to 14.7] | 10.5 [4.9 to 18.9]

ADVERSE EVENTS:
Time Frame: Day of endometrial transformation (Day -5) up to 12 weeks of pregnancy
Arm/Group | Crinone | Crinone® Plus Duphaston
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 4/86 | 4/86
Other Adverse Events (participants affected / at risk) | 17/86 | 14/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crinone (N=86) | Crinone® Plus Duphaston (N=86)
Decreased embryo viability (Injury, poisoning and procedural complications) | 2 | 2
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crinone (N=86) | Crinone® Plus Duphaston (N=86)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 8 | 4
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 | 3
Vaginal haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03858049/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03858049/SAP_001.pdf